CLINICAL TRIAL: NCT06015165
Title: Outcomes for Anesthesiologist-Led Care of Analgesic Protocol in Anorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Li Fang Wang, attending doctor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaJapanFHAnesth3
Record Dates: First submitted 2023-08-17; First posted 2023-08-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
Keywords: ambulatory surgery; anorectal surgery; postoperative analgesia; anesthesiologist-led care
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients undergoing complex anorectal surgery under general anesthesia will be included in this study. In Anes Group, the anesthesiologist routinely works in the operating room, and will communicate with anorectal physicians through bedside visits, video telephone calls, and a hospital-wide electronic medical record system in the operating room. Anesthesiologists will administer opioids or non-opioids at the optimal interval and standard dose until discharge. The anesthesiologist and the surgeon will jointly formulate the discharge medication plan and give the patient guidance on analgesic treatment. Patients in the Surg. Group will be given local anesthesia during the operation, and will receive routine ambulatory surgery anesthesia plan, and routine postoperative analgesia plan in the ward will be given to the patients, under the guidance of the department of pharmacy. The patients will receive rescue opioids and standardized NSAIDs until discharge.
Masking Description: This is an open label trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anes Group (Experimental): In Anes Group, the anesthesiologist routinely works in the operating room, and will communicate with anorectal physicians through bedside visits, video telephone calls, and a hospital-wide electronic medical record system in the operating room. Anesthesiologists will evaluate the patient's pain degree and symptoms perioperatively at bedside, and will administer opioids or non-opioids at the optimal interval and standard dose until discharge. The anesthesiologist and the surgeon will jointly formulate the discharge medication plan and give the patient guidance on analgesic treatment.
  Interventions: Drug: Analgesia plan for Anes. Group; Procedure: Multi-modal analgesia during the surgery
- Surg. group (Active Comparator): According to the current perioperative management mode, patients in the surgeon-led group (Surg. group) will be given local anesthesia during the operation, and will receive routine ambulatory surgery anesthesia plan, and routine postoperative analgesia plan in the ward will be given to the patients, under the guidance of the department of pharmacy. The patients will receive rescue opioids and standardized NSAIDs until discharge.
  Interventions: Drug: Analgesia plan for Surg. Group; Procedure: Multi-modal analgesia during the surgery

INTERVENTIONS:
Drug: Analgesia plan for Anes. Group — For Anes. Group, hydromorphone intravenous pump (PCIA) with 0.04mg/hr and 0.2mg/hr bolus controlled administration. Rescue opioids will be given as sufentanil 5μg/hr, depending on the time of the last intraoperative administration. NSAIDs such as flurbiprofen axetil or ibuprofen will be administered as a complementary treatment option.
  Other Names: Anes Group
  Arms: Anes Group
Drug: Analgesia plan for Surg. Group — For Surg. Group, hydromorphone intravenous pump is set with the same analgesic formula as in Anes. Group. Routine prescriptions for rescue opioids (tramadol) and NSAIDs according to pain level recommended by the pharmacy department will be administered.
  Other Names: Surg. Group
  Arms: Surg. group
Procedure: Multi-modal analgesia during the surgery — Multi-modal analgesia, including intraoperative long-acting local anesthetics (ropivacaine and methylene blue), perioperative narcotic analgesics, and postoperative laxative and antibiotics. PCIA with the same analgesic formula will be applied in both groups.
  Other Names: Intraoperative analgesic plan

SUMMARY:
This will be an open, prospective, parallel-group, randomized controlled trial. Patients scheduled for complex anorectal surgery under general anesthesia will be enrolled, and the perioperative analgesia mode led by anesthesiologists will be established. Compared with the perioperative analgesia mode led by surgeons, the efficacy and safety of analgesia, quality of life and satisfaction of patients will be evaluated. This study is aimed at the feasibility and efficiacy of anesthesiologist-led treatment mode in the management of moderate and severe pain in patients after complex anorectal surgery.

DETAILED DESCRIPTION:
Patients suffer from moderate to severe postoperative pain up to 14 days after anorectal surgery. To establish an anesthesiologist-led multidisciplinary team for postoperative analgesia in anorectal surgery under short and complex general anesthesia. However, the implementation of perioperative analgesia in anorectal surgery has not been paid enough attention. This study aims to establish the application of anesthesiologist-led multidisciplinary postoperative analgesia in anorectal surgery under general anesthesia.

Objectives: Patients undergoing complex anorectal surgery under general anesthesia will be randomly divided into two groups: anesthesiologist-led group (Anes Group) and surgeon-led group (Surg Group).

Interventions: Both groups will receive general anesthesia combined with long-term local anesthesia, postoperative patient controlled intravenous analgesia (PCIA) and multi-mode analgesia including laxatives and antibiotics. In Anes Group, patients receive postoperative analgesia following the protocol established by the anesthesiologist, continuous with intraoperative analgesic protocol. In Surg Group, patients will be given postoperative analgesia and follow-ups by the traditional mode formulated by the surgeons and the consultant of the pharmacists. The postoperative PCIA analgesic formula and the choice of analgesics are same in the two groups.

Follow-ups and outcomes: Patients will be followed-up till total recovery after surgery. Primary outcome is the time of recovery of work and life after surgery day, defined as not requiring any additional medication and resuming full pre-operative work life content. Secondary outcomes include opioid use after surgery, the degree of pain during defecation and rest pain, the adverse reactions related to analgesia, satisfaction, the time of ambulation, the length of hospital stay.

The purpose of this study was to evaluate the feasibility of anesthesiologist-led care model in complex anorectal surgery and to optimize the perioperative analgesia in anorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesia (ASA) grading I-III
2. ≥18 years old
3. Patients scheduled for complex anorectal surgery under general anesthesia, e.g., mixed hemorrhoidectomy/sclerosing agent injection/ligation, radical anal fistula resection, peri-anal abscess incision and drainage

Exclusion Criteria:

1. Informed consent not obtained
2. Allergic to general anesthetics, hydromorphone, non-steroidal anti-inflammatory drugs and other related ingredients
3. Opioid abuse or pathological pain that requires long-term analgesic treatment
4. History of severe asthma attack and acute phase of asthma
5. Moderate or above ventilatory function or diffusion dysfunction
6. Liver dysfunction reached Child B grade; Renal insufficiency reached chronic kidney disease (CKD) stage IV
7. Gastric retention and paralytic ileus
8. Pregnant and lactating patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
the time of recovery of work and life after surgery day | up to 21 days
  not requiring any additional medication and resuming full pre-operative work life content

SECONDARY OUTCOMES:
postoperative rest pain | up to 21 days
  postoperative rest pain in Numeric Rating Scales (NRS) 1-10, when 0 means painless, and 10 means the highest level of unbearable pain
postoperative defecation pain | up to 21 days
  postoperative defecation pain in Numeric Rating Scales (NRS) 1-10, when 0 means painless, and 10 means the highest level of unbearable pain
adverse reactions | up to 21 days
  adverse reactions including postoperative nausea and vomiting(PONV), dizziness, respiratory depression, etc.
patients' satisfaction | up to 21 days
  patients' satisfaction self-rating 1-10
total opioid use after surgery | up to 21 days
  Total opioid use from postoperative period till the discontinuation of surgery-related therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia Li, Doctor, Study Director — China-Japan Friendship Hospital
Locations (2):
- China (2):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Department of Anesthesiology, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No